CLINICAL TRIAL: NCT01073592
Title: Comparison Between Home Macular Perimeter (FORESEE HOME) and OCT Visual Field Defects in Patients With CNV
Brief Title: Comparison Between Foresee Home and Optical Coherence Tomography (OCT) Visual Field Defects in Patients With Choroidal Neovascularization (CNV)
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: FORESEE HOME-POST-03
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Age Related Macular Degeneration
Keywords: HMP; CNV; AMD; PHP; HPHP; FORESEE HOME
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CNV patiens

SUMMARY:
The Foresee Home is used in the recent years to detect age-related macular degeneration (AMD) lesions. The device is capable of differentiation as to stages of AMD and early detection of changes including choroidal neovascularization (CNV). The Foresee Home demonstrates a high level of sensitivity and specificity as to the different stages of AMD including newly diagnosed or early detection of CNV.

The OCT may be use as well to identify choroidal neovascularization (CNV). Comparison between the two methods will allow better understanding of both devices.

The Foresee Home can use as an assessment tool for the progression and success of the treatment given to AMD lesions. Therefore, evaluation the size and the location of the treated lesions may serve as an additional tool.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* Subjects diagnosed with CNV
* Did not perform more then 4 anti- VGEF injections
* VA with habitual correction better then 6/45 in the study eye
* Ability to understand instructions
* Familiar with computer usage

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy,
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the target eye
* Participation in another study with the exclusion of AREDS study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suspected to have CNV secondary to AMD in at least one eye
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Size and location of lesions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Siegal, Prof., Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- See also: sponsor web site — http://www.notalvision.com